CLINICAL TRIAL: NCT00831831
Title: Can Safety Planning Improve Perinatal Outcomes Among Pregnant Women Exposed to Intimate Partner Violence?
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The team wasn't able to work effectively with the social worker at the site
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Foundation for Women's Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H07-02007
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Perinatal Outcomes
Keywords: perinatal; intimate partner violence; randomized controlled trial; preterm; hemorrhage; safety
MeSH Terms: conditions — Premature Birth; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Safety planning — See detailed description

SUMMARY:
OBJECTIVE: To investigate if, among women exposed to physical violence during pregnancy, does a targeted intervention consisting of safety planning and referral to community advocacy services decrease rates of adverse perinatal outcomes including antepartum hemorrhage or infection, low birthweight, and perinatal death.

DESIGN: A randomized controlled trial. SETTING: Surrey Memorial Hospital and BC Women's Hospital in British Columbia, Canada PARTICIPANTS: Pregnant women experiencing intimate partner violence MAIN OUTCOME MEASURES: We are interested in perinatal outcomes such as birth weight and preterm labour.

DATA ANALYSIS: Outcomes for women in each arm of the trial will be compared in an intention to treat analysis. Changes in risk for adverse outcomes associated with the study intervention will be estimated by the odds ratios calculated by the logistic regression model.

DETAILED DESCRIPTION:
Protocol RESEARCH PLAN

Title: Massage Therapy and Labour Outcomes: a Randomized Controlled Trial

1. Goal and Objectives The overall purpose of this project is to evaluate whether or not, among women exposed to physical violence during pregnancy, does a targeted intervention consisting of safety planning and referral to community advocacy services decrease rates of adverse perinatal outcomes including antepartum hemorrhage or infection, low birthweight, and perinatal death.

Specific Aims Our specific aim is to randomly assign women who identify as having been exposed to intimate partner violence to receive either usual care or a targeted safety planning intervention in order to study effect of safety planning on perinatal outcomes.

Research Questions

We will compare among women exposed to physical violence during pregnancy, does a targeted intervention consisting of safety planning and referral to community advocacy services decrease rates of adverse perinatal outcomes including:

1. antepartum hemorrhage
2. antepartum infection
3. low birthweight
4. perinatal death

Hypotheses We hypothesize that, among women who disclose exposure to intimate partner violence during pregnancy, those receive a targeted intervention of safety planning and referral will experience a reduction in incidence of low birthweight babies compared to those who receive standard care consisting of a resource card and the offer of referral to a social worker.

2.0 Design This is a randomized controlled trial. After providing informed, written consent, each participant will be randomly assigned to a) usual care or b) a targeted intervention program. Randomization will take place by pulling a consecutively numbered card from a box, within which a concealed allocation is written.

Study sample Our study sample will include pregnant women how indicate concern about intimate partner violence to their antenatal care providers at Surrey Memorial Hospital and BC Women's Hospital.

Study Setting The study will take place at Surrey Memorial Hospital an BC Women's Hospital in Vancouver, in British Columbia, Canada.

Recruitment During our proposed study, women who indicate to their antenatal provider that they are concerned about violence will be asked if they would like to receive some information about a study related to women's safety during pregnancy. If women are agreeable, the caregiver will provide them with a recruitment brochure. Women will sign their name on this brochure if they are interested and indicate how they would like to be contacted. A study research assistant will contact potential participants in a way that they have indicated is safe, and explain the study in detail.

Randomization Randomization will take place immediately after obtaining written consent. A statistical software package (SPSS - Statistical Program for the Social Sciences) will be utilized to randomly assign sequential numbers to one of the two treatment arms. Cards will be numbered sequentially and labelled with the treatment allocation. These cards will be placed in opaque envelopes in a box which will be kept in a locked cupboard to which the recruitment nurse holds the key. Envelopes will be opened in sequential order for each study participant after written informed consent has been obtained. A log book will be maintained by the research assistant detailing the patients approached, their decision to participate or not, randomization number, and allocation.

Protocol Usual care will consist of a resource card providing information about a variety of community agencies that support women, including women experiencing violence. and the opportunity to meet with a hospital social worker for referral to relevant community agencies.

The intervention program be provided by community health nurses and will consist of:

i) ensuring that the woman has telephone numbers for community agencies serving women who experience violence, in particular, agencies that serve women of their cultural background with language-specific services; ii) knowledge of how to contact a women's shelter, and if desired, assistance in contacting the shelter and negotiating admission; iii) offer of referral to a hospital social worker with translation services available if necessary; iv) information on Canadian law with respect to violence perpetrated by an intimate partner; v) information on how to access outreach support to apply for welfare and/or skills assessment and retraining; vi) information on how to access outreach support to access emergency funds from a provincial employment and assistance program vii) safety planning, including a) identification of a method of escape from the home (a "rescue" driver, call to a shelter, taxi, extra set of car keys for family car); b) an "escape bundle" kept outside the home including important documents, money, etc.; c) identification of an escape route out of the house (unlatched window, for example); and d) recruitment of a friend or neighbour who can come over in the event that a code word is used over the phone.

Women will be asked to complete two measures of violence exposure at the time of enrollment and on a monthly basis thereafter.

Study Outcomes Our study outcomes include pregnancy complications and newborn outcomes. Pregnancy complications will include hemorrhage during the 2nd or 3rd trimester of pregnancy, intrauterine growth restriction, preterm labour (prior to 37 weeks), preterm delivery, and chorioamnionitis (infection of the placenta and membranes). Our primary newborn outcome is low birthweight (less than 2500g). Low birthweight will be further subdivided into preterm birth and/or birthweight within the 10th percentile for gestational age and sex by provincial standards. We will also document perinatal death.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Women
* Experiencing intimate partner violence
* Able to speak English or Punjabi.

Exclusion Criteria:

* None

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intrauterine Growth Restriction. | During pregnancy

SECONDARY OUTCOMES:
Hemorrhage during the 2nd or 3rd trimester of pregnancy, preterm labour, preterm delivery, and chorioamnionitis. | During pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Patti Janssen, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Surrey Memorial Hospital, Surrey, British Columbia, Canada